CLINICAL TRIAL: NCT05970471
Title: Preferences of Patients Treated With Oral Cancer Drugs and Informal Caregivers for Pharmaceutical Consultation in Hospital: Discrete Choice Method to Inform Decision-making by Healthcare Professionals
Brief Title: Preferences of Patients Treated With Oral Cancer Drugs and Informal Caregivers for Pharmaceutical Consultation in Hospital
Acronym: IMPLICATION
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/790
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Preference, Patient; Pharmacist-Patient Relations; Caregiver; Cancer
Keywords: Preference, Patient; Pharmacist-Patient Relations; Cancer of Colon; Cancer, Breast; Lung Cancer; Prostate Cancer; Renal Cancer; caregiver
MeSH Terms: conditions — Patient Preference; Neoplasms; Colonic Neoplasms; Breast Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To ensure the safe use of oral anticancer drugs, oncology pharmacy consultations (OPCs) have been established in France. Their goal is to provide the patient with the means to identify, prevent and limit adverse effects and to know who to refer to in case of a serious adverse effect, perform a pharmaceutical analysis of the prescription, and participate in the improvement and evaluation of overall compliance. OPCs are conditioned by the needs, expectations, and involvement of the patients in their care. In healthcare, patients are increasingly encouraged to play an active role in the knowledge and management of their health, express their concerns and preferences, and participate in medical decisions. Thus, it is essential to elicit their preferences. The discrete-choice experiment (DCE) is the validated and recommended method of the International Society for Pharmacoeconomics and Outcomes Research for such a task.

DETAILED DESCRIPTION:
To ensure the safe use of oral anticancer drugs, oncology pharmacy consultations (OPCs) have been established in France. Their goal is to provide the patient with the means to identify, prevent and limit adverse effects and to know who to refer to in case of a serious adverse effect, perform a pharmaceutical analysis of the prescription, and participate in the improvement and evaluation of overall compliance. OPCs are conditioned by the needs, expectations, and involvement of the patients in their care. In healthcare, patients are increasingly encouraged to play an active role in the knowledge and management of their health, express their concerns and preferences, and participate in medical decisions. Thus, it is essential to elicit their preferences. The discrete-choice experiment (DCE) is the validated and recommended method of the International Society for Pharmacoeconomics and Outcomes Research for such a task.

ELIGIBILITY:
of patients:

Main inclusion Criteria:

* Patients with lung, prostate breast, prostate or renal cancer;
* Patients with oral cancer drugs;
* Patients accepted to take par in pharmaceutical consultation in hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 240 patients - 60 Caregivers - 360 healhcare professionnals (pharmacist, oncologists, general practitioners)
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-12-04 (Actual); Study Completion 2025-12-04 (Actual)

PRIMARY OUTCOMES:
Preferences of patients | 12 months
  utility associated with each attribute

SECONDARY OUTCOMES:
Preferences of cargivers and healthcare profesionnals | 12 months
  utility associated with each attribute

CONTACTS AND LOCATIONS:
Overall Officials: Virginie NERICH, PhD, Principal Investigator — CHU de Besançon
Locations (1):
- CHU de Besançon, Besançon, France